CLINICAL TRIAL: NCT03692195
Title: Assessment of Sleep by WHOOP in Ambulatory Subjects
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Arizona (Other)
Collaborators: Whoop Inc. (Industry)
Responsible Party: Principal Investigator, Sairam Parthasarathy, Professor of Medicine, University of Arizona
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Other
Other Study IDs: WHOOP00001
Record Dates: First submitted 2018-09-27; First posted 2018-10-02 (Actual); Last update posted 2021-08-09 (Actual); Status verified 2021-08

CONDITIONS: Sleep Quality
Keywords: sleep; healthy volunteers; sleep study
MeSH Terms: conditions — Sleep Initiation and Maintenance Disorders

STUDY DESIGN:
Intervention Model Description: Study participants will either wear the WHOOP strap 2.0 one week before their sleep study (as well as the night of the sleep study) or one week after their sleep study (as well as the night of the sleep study). This is a within subjects design to compare sleep patterns the week subjects are wearing the Whoop strap 2.0 with the week subjects do not wear the Whoop Strap 2.0. Participants either wear the WHOOP strap 2.0 one week before or one week after their sleep study in order to counterbalance for ordering effects.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Week WHOOP is worn (Experimental): Participants will wear the WHOOP strap 2.0 either 7 days prior to or 7 days after their sleep study.
  Interventions: Device: WHOOP Strap 2.0
- Week WHOOP is not worn (Placebo Comparator): Participants will not wear the WHOOP strap 2.0 either 7 days prior to or 7 days after their sleep study.
  Interventions: Other: No Device

INTERVENTIONS:
Device: WHOOP Strap 2.0 — The WHOOP Strap 2.0 is worn on the wrist, continuously throughout the 7-day period of which participants will be assigned. It measures heart rate, sleep, strain, and recovery.
  Arms: Week WHOOP is worn
Other: No Device — The WHOOP Strap 2.0 is not worn on the wrist for a seven day period.
  Arms: Week WHOOP is not worn

SUMMARY:
Polysomnography (PSG) is considered the 'gold standard' for objectively measuring different parameters of sleep, including total sleep time, quality of sleep, and distinguishing between sleep stages. However, PSG is costly, and tends to be burdensome in terms of set-up time and invasiveness during sleep. Wearable sleep-monitoring devices could prove to be a more practical alternative to PSG.

Additionally, while EKG leads are typically what is utilized to measure heart rate (HR) and heart rate variability (HRV) throughout the night in a PSG set-up, every day-use HR monitors are also beneficial for individuals to evaluate their cardiovascular activity during different types of physical activities (including every day activities, exercise, and sleep), as well as their heart's ability to "recover" from a given activity.

The investigators propose to study the effect of the WHOOP Strap 2.0 device on sleep perception and perform a methodological study to validate the accuracy of the the WHOOP Strap 2.0 device when measuring HR accuracy and HRV accuracy, and sleep quality and quantity with respect to PSG in healthy volunteers with no self-reported sleep disorders or debilitating medical conditions.

DETAILED DESCRIPTION:
Polysomnography (PSG) is still considered the 'gold standard' for measuring sleep parameters, such as total sleep time, sleep efficiency, and sleep stages (6). However, PSG suffers from key limiting factors for routine care applications irrespective of setting (e.g., home, acute setting, and long term setting). Some of the key limitations of PSG are the high cost, arduous application, intrusiveness to sleep, and requirement of sleep lab and dedicated infrastructure. Wearable technologies could provide a viable alternative to PSG. We are proposing to perform a methodological study aimed at validating the accuracy of WHOOP Strap 2.0 to measure sleep quantity and sleep quality in ambulatory subjects. We will measure sleep by both WHOOP Strap 2.0 and PSG in healthy volunteers (age 18 - 45 years) without self-reported sleep disorders or chronic disabling medical conditions.

In ambulatory patients, sleep is usually assessed by the American Academy of Sleep Medicine guidelines which derives from the Rechtschaffen and Kales (R&K) method with good to excellent inter-observer reliability for assessing sleep in the same population; but the Cohen's K range is still 0.68 to 0.82 and much lower for non rapid eye movement (NREM) sleep stage 1 (N1). To account for such inter- and intra-rater reliability issues with the PSG gold-standard, we will only consider sleep stages that are unequivocally scored as a particular stage (light NREM, slow wave sleep [SWS] or REM sleep [R sleep]) by two different observers.

Additionally, while there are many devices available to healthy individuals to measure heart rate, there aren't many available that provide a daily heart rate variability statistic. Heart rate variability can be defined as the variation over time of the period between consecutive heart beats. This is due to the balancing regulation effects of the parasympathetic (PNS) and sympathetic (SNS) actions of the autonomic nervous system (ANS). Increased SNS action results in a "fight or flight" response, leading to an accelerated heart rate, while increased PNS activity results in a "rest and digest" response, leading to a decelerated heart rate. The increased variability of heart rate (HR) is an indication of the ANS' control on HR and the heart's ability to respond. WHOOP Strap 2.0 provides users with real-time HR and a daily HRV statistic that is included in other variables calculated measuring daily strain and recovery statistics. We will measure HR and HRV by both WHOOP Strap 2.0 and EKG leads in healthy volunteers (ages 18-45 years) without chronic disabling medical conditions.

ELIGIBILITY:
Inclusion Criteria:

* Ability to provide informed consent
* Willingness to undergo a polysomnography electrode hook-up and wear a WHOOP strap 2.0.
* Healthy volunteers

Exclusion Criteria:

* Presence of untreated sleep disorder that requires diagnostic testing and treatment (insomnia, obstructive sleep apnea, narcolepsy, restless leg syndrome, REM sleep behavior disorder, or circadian rhythm sleep disorders).
* Apnea-Hypopnea index greater than or equal to 15 per hour as per AASM guidelines
* Active substance abuse or alcoholism
* Pregnancy or lactation
* Currently taking sedative medications
* Chronic medical conditions such as hypertension, diabetes mellitus, cardiac disorders, arthritis, or other chronic medical conditions
* BMI greater than 26

Ages: 18 Years to 45 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 35 (Actual)
Dates: Start 2018-11-01 (Actual); Primary Completion 2019-06-07 (Actual); Study Completion 2019-06-07 (Actual)

PRIMARY OUTCOMES:
PROMIS Sleep Questionnaire Short Form | Baseline, Day 7, and Day 14 (~2 weeks)
  An 8-item questionnaire used to assess subjective sleep disturbance in individuals 18 and older. Each questionnaire item addresses an aspect about sleep quality that is rated by the respondent on a 5-point scale (i.e., 1= Not at all & 5 = Very Much). Change in PROMIS score will be assessed between Baseline, Day 7, and Day 14.

SECONDARY OUTCOMES:
Sleep duration by WHOOP Strap 2.0 | The WHOOP Strap 2.0 is worn on day 7 of the study. Polysomnography occurs on day 7 of the study.
  Sleep duration is defined as the amount of time one spends asleep. This is measured by the WHOOP Strap 2.0 and is compared to Polysomnography, the gold standard for measuring sleep parameters and sleep stages.
Sleep Fragmentation | The WHOOP Strap 2.0 is worn on day 7 of the study. Polysomnography occurs on day 7 of the study.
  Sleep fragmentation is defined as interruptions in sleep. This is measured by the WHOOP Strap 2.0 and is compared to Polysomnography, the gold standard for measuring sleep parameters and sleep stages.
Heart Rate Variability | The WHOOP strap 2.0 is worn continuously throughout the duration of the study (~14 days).
  Heart Rate Variability is defined as the physiological phenomenon of the variation of time intervals between heart beats. This will be measured by the WHOOP Strap 2.0.
Sleep Staging | The WHOOP Strap 2.0 is worn on day 7 of the study. Polysomnography occurs on day 7 of the study.
  The WHOOP Strap 2.0 differentiates between light sleep, slow wave sleep, and REM sleep. This will be compared to polysomnography, which is the gold standard of measuring sleep staging and sleep parameters.
Sleep Versus Wake Detection | The WHOOP Strap 2.0 is worn on day 7 of the study. Polysomnography occurs on day 7 of the study.
  The WHOOP Strap 2.0 differentiates between sleep and wake status. This will be compared to polysomnography, which is the gold standard of measuring sleep staging and sleep parameters.
Heart Rate Accuracy | The WHOOP Strap 2.0 is worn on day 7 of the study. Polysomnography occurs on day 7 of the study.
  The WHOOP Strap 2.0 collects heart rate. This will be compared to the known gold standard of Electrocardiogram electrode leads as part of the polysomnography montage.
Respiratory Rate | The WHOOP Strap 2.0 is worn on day 7 of the study. Polysomnography occurs on day 7 of the study.
  The WHOOP Strap 2.0 collects respiratory rate. This will be compared to the nasal cannula respiratory rate which is part of the polysomnography montage.

CONTACTS AND LOCATIONS:
Overall Officials: Sairam Parthasarathy, MD, Principal Investigator — University of Arizona
Locations (1):
- Center for Sleep and Circadian Sciences, Tucson, Arizona, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Berryhill S, Morton CJ, Dean A, Berryhill A, Provencio-Dean N, Patel SI, Estep L, Combs D, Mashaqi S, Gerald LB, Krishnan JA, Parthasarathy S. Effect of wearables on sleep in healthy individuals: a randomized crossover trial and validation study. J Clin Sleep Med. 2020 May 15;16(5):775-783. doi: 10.5664/jcsm.8356. Epub 2020 Feb 11. PMID 32043961